CLINICAL TRIAL: NCT02414282
Title: F 18 T807 Tau PET Imaging of Progressive Posterior Cortical Dysfunction Due to Alzheimer Disease
Brief Title: F 18 T807 Tau PET Imaging of Progressive Posterior Cortical Dysfunction (IND 123119, Protocol E)
Acronym: Protocol E
Status: Completed | Type: Observational
Sponsor: Tammie L. S. Benzinger, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, Tammie L. S. Benzinger, MD, PhD, Professor of Radiology & Neurological Surgery, Washington University School of Medicine
Organization: Washington University School of Medicine (Other)
Other Study IDs: IND 123119 Protocol E
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2021-01-19 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer Disease; Progressive Posterior Cortical Dysfunction (PPCD)
Keywords: Dementia; Brain Diseases; mild cognitive impairment; Central Nervous System Diseases; Neurodegenerative Disease
MeSH Terms: conditions — Alzheimer Disease; Dementia; Brain Diseases; Cognitive Dysfunction; Central Nervous System Diseases; Neurodegenerative Diseases | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Experimental F 18 T807
  Interventions: Drug: F 18 T807

INTERVENTIONS:
Drug: F 18 T807 — Participants will receive a single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807. For those who cannot tolerate the full exam, participants will receive single intravenous bolus injection of approximately 6.5-10mCi (240-370MBq) of F 18 T807.
  Other Names: 18F-AV-1451

SUMMARY:
This project will collect quantitative pilot data that will allow the characterization of uptake and binding of 18F-AV-1451 (also known as F 18 T807), a novel tau imaging compound, in individuals with Progressive Posterior Cortical Dysfunction (PPCD) and logopenic variant primary progressive aphasia (lvPPA). The primary goal is to develop tau imaging technique as an antecedent biomarker of cognitive decline. The investigators propose to obtain preliminary data that will support the possibility of detecting cognitive decline in its earliest stages, before the occurrence of dementia.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants, at least 45 years of age.
2. Clinical diagnosis of PPCD.
3. Participant is able and willing to undergo testing (MRI or CT, PET, radioactive tracer injection, LP; for those unable to undergo an MRI, CT will be used to generate regions-of-interest).
4. Pre-menopausal women will have a negative urine pregnancy test within 24 hours of T807 drug administration.

Exclusion Criteria:

1. Has any condition that, in the Investigator's opinion, could increase risk to the participant, limit the participant's ability to tolerate the experimental procedures, or interfere with the collection/analysis of the data (for example, participants with severe chronic back pain might not be able to lie still during the scanning procedures).
2. Is deemed likely unable to perform the imaging procedures for any reason.
3. Has a high risk for Torsades de Pointes or is taking medications known to prolong QT interval.
4. Has hypersensitivity to F 18 T807 or any of its excipients.
5. Contraindications to PET, PET-CT or MR (e.g. electronic medical devices, inability to lie still for long periods) that make it unsafe for the individual to participate.
6. Severe claustrophobia.
7. Currently pregnant or breast-feeding.
8. For those electing to undergo the optional lumbar puncture: on anticoagulant of any form prior to lumbar puncture.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Collaborating physicians and the Knight ADRC Clinical Core will refer participants to the Knight ADRC Research Imaging (KARI) Program for MR and PET imaging to evaluate tau distribution in the brains of cognitively normal and cognitively impaired individuals, with the primary goal of developing this highly promising tau imaging technique as an antecedent biomarker of cognitive decline. We propose to recruit groups of patients with PPCD and lvPPA from the same clinical environment.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-10-20 (Actual); Study Completion 2020-10-20 (Actual)

PRIMARY OUTCOMES:
F 18 T807 Standard Uptake Value Ratios (SUVR) will be correlated with other imaging modalities (MRI, PET amyloid imaging) and cognitive performance. | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Tammie Benzinger, MD, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
We will share this data with other researchers. They may be doing research in areas similar to this research or in other unrelated areas. These researchers may be at Washington University, at other research centers and institutions, or industry sponsors of research. We may also share your research data with large data repositories (a repository is a database of information) for broad sharing with the research community. If the individual research data is placed in one of these repositories only qualified researchers, who have received prior approval from individuals that monitor the use of the data, will be able to look at the information.

REFERENCES:
- [Result] Day GS, Gordon BA, Jackson K, Christensen JJ, Rosana Ponisio M, Su Y, Ances BM, Benzinger TLS, Morris JC. Tau-PET Binding Distinguishes Patients With Early-stage Posterior Cortical Atrophy From Amnestic Alzheimer Disease Dementia. Alzheimer Dis Assoc Disord. 2017 Apr-Jun;31(2):87-93. doi: 10.1097/WAD.0000000000000196. PMID 28394771